CLINICAL TRIAL: NCT00289185
Title: A Phase IIb Randomized, Double-blind, Controlled Study of the Safety, Immunogenicity and Proof-of-concept of RTS,S/AS02D, a Candidate Malaria Vaccine, When Incorporated Into an Expanded Program on Immunization (EPI) Regimen That Includes DTPw/Hib in Infants Living in a Malaria-endemic Region.
Brief Title: Study of Safety, Immunogenicity and Efficacy of a Candidate Malaria Vaccine in Tanzanian Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 104298; 2015-001539-19 (EudraCT Number)
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Malaria; Malaria Vaccines
Keywords: Coccidiosis; Parasitic Diseases; Malaria, Falciparum; Malaria
MeSH Terms: conditions — Malaria; Coccidiosis; Parasitic Diseases; Malaria, Falciparum | interventions — RTS malaria vaccine; Engerix-B

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- RTS,S/AS02D Group (Experimental): Subjects aged between 6 and 10 weeks at the time of first vaccination received by intramuscular injection a 3-dose vaccination course of the RTS,S/AS02D vaccine co-administered with the TETRActHib™ vaccine at Week 0, Week 4 (Month 1) and Week 8 (Month 2). The RTS,S/AS02D vaccine was administered in the left anterolateral thigh, and the TETRActHib™ vaccine in the right anterolateral thigh.
  Interventions: Biological: RTS,S/AS02D; Biological: TETRActHib™
- Engerix-B Group (Active Comparator): Subjects aged between 6 and 10 weeks at the time of first vaccination received by intramuscular injection a 3-dose vaccination course of Engerix-B® vaccine co-administered with the TETRActHib™ vaccine at Week 0, Week 4 (Month 1) and Week 8 (Month 2). The Engerix-B® vaccine was administered in the left anterolateral thigh, and the TETRActHib™ vaccine in the right anterolateral thigh..
  Interventions: Biological: Engerix-B®; Biological: TETRActHib™

INTERVENTIONS:
Biological: RTS,S/AS02D — 3-dose intramuscular injection in the thigh
  Other Names: GSK 257146; RTS; S/AS02D
  Arms: RTS,S/AS02D Group
Biological: Engerix-B® — 3-dose intramuscular injection in the thigh.
  Arms: Engerix-B Group
Biological: TETRActHib™ — 3-dose intramuscular injection in the thigh.
  Other Names: DTPw/Hib

SUMMARY:
GSK Biologicals in partnership with the Malaria Vaccine Initiative at PATH is developing a candidate malaria vaccine GSK 257049 for the routine immunization of infants and children living in malaria endemic areas. The vaccine would offer protection against malaria disease due to the parasite Plasmodium falciparum. The vaccine would also provide protection against infection with hepatitis B virus (HBV).

In order to integrate the malaria vaccine into the EPI regimen in malaria-endemic regions, a new variant RTS,S/AS02D (0.5 mL dose) has been developed.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
This is a phase 2b trial designed to evaluate the safety and immunogenicity of RTS,S/AS02D when co-administered with a multivalent DTPw/Hib (Aventis Pasteur's TETRActHib vaccine). Infants randomized to the control group will receive a licensed hepatitis B vaccine, Engerix-B in place of RTS,S/AS02D.

Data pertaining to RTS,S/AS02D or Engerix-B will be collected in a double blinded manner; data relating to TETRActHib will be collected in an open fashion.

Oral polio vaccine (OPV) will be administered at birth, 8, 12, 16 weeks in co-administration with other vaccines and will not be administered as part of this protocol. Antibody titers to OPV will not be assessed as part of this protocol.

ELIGIBILITY:
Inclusion criteria:

* A male or female infant between 6 and 10 weeks of age at the time of first vaccination.
* Written or oral, signed or thumb-printed and witnessed informed consent obtained from the parent(s)/guardian(s) of the child.
* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol (e.g. return for follow-up visits).
* Born to a mother who is HBsAg negative & HIV negative.
* Born after a normal gestation period (between 36 and 42 weeks).
* Subjects who live within a 5 km radius of a dispensary.

Exclusion criteria:

* Acute disease at the time of enrolment.
* Serious acute or chronic illness determined by clinical or physical examination and laboratory screening tests.
* Laboratory screening tests out of range for haemoglobin, total white cell count, platelets, ALT and creatinine.
* Previous vaccination with diphtheria, tetanus, pertussis (whole-cell or acellular), Hemophilus influenzae type b or hepatitis B vaccines.
* BCG administration within one week of proposed administration of a study vaccine.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine(s).
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of immunoglobulins, blood transfusions or other blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Previous participation in any other malaria vaccine trial.
* Simultaneous participation in any other clinical trial.
* Same sex twin.
* Maternal death.
* History of allergic reactions (significant IgE-mediated events) or anaphylaxis to previous immunizations.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 340 (Actual)
Dates: Start 2006-09-27 (Actual); Primary Completion 2008-02-11 (Actual); Study Completion 2009-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Abdulla S, Oberholzer R, Juma O, Kubhoja S, Machera F, Membi C, Omari S, Urassa A, Mshinda H, Jumanne A, Salim N, Shomari M, Aebi T, Schellenberg DM, Carter T, Villafana T, Demoitie MA, Dubois MC, Leach A, Lievens M, Vekemans J, Cohen J, Ballou WR, Tanner M. Safety and immunogenicity of RTS,S/AS02D malaria vaccine in infants. N Engl J Med. 2008 Dec 11;359(24):2533-44. doi: 10.1056/NEJMoa0807773. Epub 2008 Dec 8. PMID 19064623
- [Derived] Abdulla S, Salim N, Machera F, Kamata R, Juma O, Shomari M, Kubhoja S, Mohammed A, Mwangoka G, Aebi T, Mshinda H, Schellenberg D, Carter T, Villafana T, Dubois MC, Leach A, Lievens M, Vekemans J, Cohen J, Ballou WR, Tanner M. Randomized, controlled trial of the long term safety, immunogenicity and efficacy of RTS,S/AS02(D) malaria vaccine in infants living in a malaria-endemic region. Malar J. 2013 Jan 8;12:11. doi: 10.1186/1475-2875-12-11. PMID 23297680
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 104298 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104298 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104298 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104298 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104298 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104298 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 340 subjects were enrolled for this study. The study comprised 2 phases, a double-blind phase, from Week 0 to Month 9 (2 months after the administration of the last vaccine dose), followed by a single-blind safety phase, from Month 9 to study end at Month 20.
Groups:
- Engerix-B Group: Subjects aged between 6 and 10 weeks at the time of first vaccination received by intramuscular injection a 3-dose vaccination course of Engerix-B® vaccine co-administered with the TETRActHib™ vaccine at Week 0, Week 4 (Month 1) and Week 8 (Month 2). The Engerix-B vaccine was administered in the left anterolateral thigh, and the TETRActHib™ vaccine in the right anterolateral thigh.
Period: Overall Study
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Started | 170 | 170
Completed | 142 | 144
Not Completed | 28 | 26
Not completed — Withdrawal by Subject | 4 | 8
Not completed — Lost to Follow-up | 23 | 17
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engerix-B Group | RTS,S/AS02D Group | Total
Number analyzed (Participants) | 170 | 170 | 340
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 7.87 (0.83) | 7.82 (0.77) | 7.85 (0.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 91 | 176
  Male | 85 | 79 | 164

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Antibodies Against Hepatitis B (Anti-HB)
Description: Concentrations were expressed as geometric mean concentrations (GMCs) in milli-international unit per milliliter (mIU/mL). The cut-off of the assay was the seroprotection cut-off of 10 mIU/mL. Month 3 results are the specific results for this primary outcome measure.
Time Frame: Prior to vaccination at Week 0 (PRE), at Month 2 and at Month 3.
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity, which included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity outcome variables were available.
Measure: Geometric Mean (95% Confidence Interval); unit: milli-international unit per milliliter
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 148 | 149
milli-international unit per milliliter
  Anti-HB - PRE (N=134;116) | 13.0 [9.8 to 17.2] | 14.3 [10.8 to 19.0]
  Anti-HB - Month 2 (N=148;149) | 16.9 [13.5 to 21.2] | 111.8 [89.9 to 139.0]
  Anti-HB - Month 3 (N=141;141) | 113.8 [91.3 to 141.8] | 667.4 [533.8 to 834.4]

2. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Week 0 to Month 9.
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subject
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 170 | 170
Subject | 42 | 31

3. Primary Outcome: Concentrations of Antibodies Against Diphtheria (Anti-D)
Description: Antibodies were measured by Enzyme-linked immunosorbent assay (ELISA). Concentrations were expressed as geometric mean concentrations (GMCs) in international unit per milliliter (IU/mL). The cut-off of the assay was the seroprotection cut-off of 0.1 IU/mL. Month 3 results are the specific results for this primary outcome measure.
Time Frame: Prior to vaccination at Week 0 (PRE), and at Month 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: international unit per milliliter
Groups:
- RTS,S/AS02D Group: Subjects aged between 6 and 10 weeks at the time of first vaccination received by intramuscular injection a 3-dose vaccination course of the RTS,S/AS02D vaccine co-administered with the TETRActHib vaccine at Week 0, Week 4 (Month 1) and Week 8 (Month 2). The RTS,S/AS02D vaccine was administered in left anterolateral thigh, and the TETRActHib vaccine in the right anterolateral thigh.
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 165 | 162
international unit per milliliter
  Anti-D - PRE (N=165;162) | NA [NA to NA] — GMC for this time point was not computed as concentrations fell below the seroprotection cut-off of 0.1 IU/mL. | NA [NA to NA] — GMC for this time point was not computed as concentrations fell below the seroprotection cut-off of 0.1 IU/mL
  Anti-D - Month 3 (N=151;149) | 1.3 [1.1 to 1.5] | 1.1 [1.0 to 1.3]

4. Primary Outcome: Concentrations of Antibodies Against Tetanus (Anti-T)
Description: as for outcome 3
Time Frame: Prior to vaccination at Week 0 (PRE), and at Month 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: international unit per milliliter
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 165 | 162
international unit per milliliter
  Anti-T - PRE (N=165;162) | 1.1 [0.9 to 1.4] | 1.2 [1.0 to 1.6]
  Anti-T - Month 3 (N=151;149) | 4.2 [3.6 to 4.8] | 3.0 [2.6 to 3.4]

5. Primary Outcome: Concentrations of Anti-polyribosyl Ribitol Phosphate Antibodies (Anti-PRP).
Description: Concentrations were expressed as geometric mean concentrations (GMCs) in microgram per milliliter (µg/mL). The cut-off of the assay is the seroprotection cut-off value of 0.15 µg/mL. Month 3 results are the specific results for this primary outcome measure.
Time Frame: Prior to vaccination at Week 0 (PRE), and at Month 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: international unit per milliliter
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 165 | 162
international unit per milliliter
  Anti-PRP - PRE (N=165;162) | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.2]
  Anti-PRP - Month 3 (N=151;148) | 19.3 [15.6 to 24.0] | 14.3 [11.5 to 17.9]

6. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 2
Time Frame: From Month 9 to Month 20.
Measure: Number; unit: Subject
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 170 | 170
Subject | 34 | 34

7. Primary Outcome: Concentrations of Anti-Bordetella Pertussis Toxin Antibodies (Anti-BPT).
Description: Antibodies were measured by Enzyme-linked immunosorbent assay (ELISA). Concentrations were expressed as geometric mean concentrations (GMCs) in ELISA unit per milliliter (EL.U/mL). The cut-off of the assay was the seropositivity cut-off of 15 EL.U/mL. Month 3 results are the specific results for this primary outcome measure.
Time Frame: Prior to vaccination at Week 0 (PRE), and at Month 3.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA unit per millilite
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 162 | 165
ELISA unit per millilite
  Anti-BPT - PRE (N=165;162) | 7.6 [7.4 to 7.8] | 7.6 [7.4 to 7.7]
  Anti-BPT - Month 3 (N=144;148) | 101.4 [92.5 to 111.2] | 82.3 [75.4 to 89.9]

8. Primary Outcome: Number of Subjects With Hepatitis B Antibody (Anti-HB) Concentrations Equal to or Above (>=) the Seroprotection Cut-off Value
Description: The seroprotection cut-off value was 10 milli-international units per milliliter (mIU/mL). Blood samples were collected prior to vaccination at Week 0 (PRE), at Month 2 and at Month 3. Month 3 results are the specific results for this primary outcome measure.
Time Frame: Prior to vaccination at Week 0 (PRE), at Month 2 and at Month 3.
Population: as for outcome 1
Measure: Number; unit: Subject
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 148 | 149
Subject
  Anti-HB >= 10 mIU/mL - PRE (N=134;116) | 45 | 44
  Anti-HB >= 10 mIU/mL - Month 2 (N=148;149) | 82 | 141
  Anti-HB >= 10 mIU/mL - Month 3 (N=141;141) | 133 | 141

9. Primary Outcome: Number of Subjects With Anti-diphtheria Antibody (Anti-D) Concentrations Equal to or Above (>=) the Seroprotection Cut-off Value
Description: Antibodies were measured by Enzyme-linked immunosorbent assay (ELISA). The seroprotection cut-off value was 0.1 international unit per milliliter (IU/mL). Blood samples were collected prior to vaccination at Week 0 (PRE), and at Month 3. Month 3 results are the specific results for this primary outcome measure.
Time Frame: Prior to vaccination at Week 0 (PRE), and at Month 3.
Population: as for outcome 1
Measure: Number; unit: Subject
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 165 | 162
Subject
  Anti-D >= 0.1 IU/mL - PRE (N=165;162) | 27 | 24
  Anti-D >= 0.1 IU/mL - Month 3 (N=151;149) | 148 | 148

10. Primary Outcome: Number of Subjects With Anti-tetanus Antibody (Anti-T) Concentrations Equal to or Above (>=) the Seroprotection Cut-off Value
Description: as for outcome 9
Time Frame: Prior to vaccination at Week 0 (PRE), and at Month 3.
Population: as for outcome 1
Measure: Number; unit: Subject
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 165 | 162
Subject
  Anti-T >= 0.1 IU/mL - PRE (N=165;162) | 156 | 155
  Anti-T >= 0.1 IU/mL - Month 3 (N=151;149) | 151 | 149

11. Primary Outcome: Number of Subjects With Anti-polyribosyl Ribitol Phosphate Antibody (Anti-PRP) Concentrations Equal to or Above (>=) the Seroprotection Cut-off Value
Description: Antibodies were measured by Enzyme-linked immunosorbent assay (ELISA). The seroprotection cut-off value was 0.15 microgram per milliliter (µg/mL). Blood samples were collected prior to vaccination at Week 0 (PRE), and at Month 3. Month 3 results are the specific results for this primary outcome measure.
Time Frame: Prior to vaccination at Week 0 (PRE), and at Month 3.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 165 | 162
Subjects
  Anti-PRP >= 0.15 µg/mL - PRE (N=165;162) | 86 | 78
  Anti-PRP >= 0.15 µg/mL - Month 3 (N=151;148) | 150 | 147

12. Primary Outcome: Number of Subjects With Anti-Bordetella Pertussis Toxin Antibody (Anti-BPT) Concentrations Equal to or Above (>=) the Seropositivity Cut-off Value
Description: Antibodies were measured by Enzyme-linked immunosorbent assay (ELISA). The seropositivity cut-off value was 15 ELISA units per milliliter (EL.U/mL). Blood samples were collected prior to vaccination at Week 0 (PRE), and at Month 3. Month 3 results are the specific results for this primary outcome measure.
Time Frame: Prior to vaccination at Week 0 (PRE), and at Month 3.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 165 | 162
Subjects
  Anti-BPT >= 15 EL.U/mL - PRE (N=165;162) | 2 | 1
  Anti-BPT >= 15 EL.U/mL - Month 3 (N=144;148) | 142 | 148

13. Secondary Outcome: Concentrations of Anti-Circumsporozoite Protein (Anti-CS) Antibodies
Description: Antibodies were measured by Enzyme-linked immunosorbent assay (ELISA). Concentrations are expressed as geometric mean concentrations (GMCs) in ELISA unit per milliliter (EL.U/mL). The cut-off of the assay was the seropositivity cut-off value of 0.5 EL.U/mL.
Time Frame: Prior to vaccination at Week 0 (PRE), at Month 2, at Month 3 and at Month 9.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA unit per milliliter
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 156 | 151
ELISA unit per milliliter
  Anti-CS - PRE (N=152;141) | NA [NA to NA] — GMC was not computed as concentrations fell below the seropositivity cut-off of 0.5 EL.U/mL | NA [NA to NA] — GMC was not computed as concentrations fell below the seropositivity cut-off of 0.5 EL.U/mL
  Anti-CS - Month 2 (N=156;151) | NA [NA to NA] — GMC was not computed as concentrations fell below the seropositivity cut-off of 0.5 EL.U/mL | 28.9 [22.4 to 37.3]
  Anti-CS - Month 3 (N=144;143) | NA [NA to NA] — GMC was not computed as concentrations fell below the seropositivity cut-off of 0.5 EL.U/mL | 69.5 [53.9 to 89.6]
  Anti-CS - Month 9 (N=147;143) | NA [NA to NA] — GMC was not computed as concentrations fell below the seropositivity cut-off of 0.5 EL.U/mL | 6.2 [4.6 to 8.3]

14. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain and swelling following vaccination with the RTS,S/AS02D or Engerix-B vaccine.
Time Frame: Within 7 days (Days 0-6) after vaccination with the RTS,S/AS02D or Engerix-B vaccine.
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subject
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 170 | 170
Subject
  Pain | 167 | 161
  Swelling | 17 | 19

15. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain and swelling following vaccination with the TETRActHib vaccine..
Time Frame: Within 7 days (Days 0-6) after vaccination with the TETRActHib vaccine.
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subject
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 170 | 170
Subject
  Pain | 169 | 168
  Swelling | 68 | 67

16. Secondary Outcome: Number of Subjects With Solicited General Symptoms.
Description: Assessed solicited general symptoms were drowsiness, fever, irritability, and loss of appetite. Fever was defined as axillary temperature above or equal to (>=) 37.5 degrees Celsius (°C).
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subject
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 170 | 170
Subject
  Drowsiness | 4 | 3
  Fever (Temperature ≥ 37.5°C) | 52 | 103
  Irritability | 71 | 81
  Loss of Appetite | 5 | 5

17. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs).
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 30 days (Days 0-29) after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 170 | 170
Subjects | 141 | 137

18. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 2
Time Frame: Throughout the entire study, from Week 0 to Month 20.
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 170 | 170
Subjects | 62 | 57

19. Secondary Outcome: Time to First Malaria Infection
Description: Malaria infection by Plasmodium falciparum (P. falciparum) was detected by active detection of infection (ADI) and passive case detection (PCD), and was defined as the presence of P. falciparum asexual parasitemia above 0 per microliter (µL) on Giemsa stained thick blood films. The time to first malaria infection is expressed in terms of rate of first malaria infection, that is, the number of malaria infection events reported (n) over the period elapsed until the event occurred (i.e. events per Persons Year at Risk [PYAR]) for each group.
Time Frame: Over the period starting 14 days after Dose 3 of RTS,S or HBV vaccine and extending for 6 months thereafter (from Month 2.5 up to Month 9).
Population: The analysis was performed on the According-to-Protocol cohort for efficacy, which included all evaluable subjects for whom data concerning efficacy outcome variables were available.
Measure: Number; unit: n/PYAR
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 151 | 146
n/PYAR | 0.29 | 0.12

20. Secondary Outcome: Number of Subjects Prevalent for Parasitemia
Description: Subjects prevalent for P. falciparum parasitemia were defined as subjects with the presence of P. falciparum asexual parasitemia above 0 per microliter (µL) on Giemsa stained thick blood films.
Time Frame: At Month 9
Population: as for outcome 19
Measure: Number; unit: Subjects
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Number analyzed (Participants) | 92 | 93
Subjects | 1 | 0

21. Secondary Outcome: Plasmodium Falciparum (P. Falciparum) Parasite Density in Subjects Prevalent for Parasitemia
Description: The parasite density in subjects prevalent for P. falciparum parasitemia (Subjects with the presence of P. falciparum asexual parasitemia above 0 per microliter (µL) on Giemsa stained thick blood films), was detected at a cross sectional time point 7 months after administration of Dose 3 of RTS,S or HBV vaccine (Month 9). Parasite density is expressed as mean, minimum and maximum density in parasite per µL. This outcome for solely assessed in the Engerix-B Group, as no subject in the RTS,S/AS02D was assessed as prevalent for parasitemia.
Time Frame: At Month 9
Population: as for outcome 19
Measure: Mean (Full Range); unit: Parasite per microliter (µL)
Arm/Group | Engerix-B Group
Number analyzed (Participants) | 1
Parasite per microliter (µL) | 23276 [23276 to 23276]

ADVERSE EVENTS:
Time Frame: Time frames for adverse events (AEs) reporting were the 7-day (Days 0-6) and 21-day (Days 0-20) periods post vaccination for solicited symptoms and unsolicited AES, respectively. Serious adverse events were assessed throughout, from Week 0 to Month 20.
Arm/Group | Engerix-B Group | RTS,S/AS02D Group
Serious Adverse Events (participants affected / at risk) | 62/170 | 57/170
Other Adverse Events (participants affected / at risk) | 169/170 | 170/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Engerix-B Group (N=170) | RTS,S/AS02D Group (N=170)
Anaemia (Blood and lymphatic system disorders) | 16 | 16
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 3
Pyrexia (General disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Abscess (Infections and infestations) | 2 | 2
Abscess limb (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0
Acarodermatitis (Infections and infestations) | 2 | 0
Bronchiolitis (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 1 | 0
Cerebral malaria (Infections and infestations) | 0 | 1
Dysentery (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 12 | 16
Malaria (Infections and infestations) | 1 | 0
Measles (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 1
Plasmodium falciparum infection (Infections and infestations) | 25 | 19
Pneumonia (Infections and infestations) | 36 | 25
Pneumonia viral (Infections and infestations) | 2 | 0
Pyoderma (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 3 | 4
Viral infection (Infections and infestations) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 2
Febrile convulsion (Nervous system disorders) | 2 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Loeffler's syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary pneumatocele (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Engerix-B Group (N=170) | RTS,S/AS02D Group (N=170)
Pain (General disorders) | 169 | 168
Swelling (General disorders) | 68 | 67
Fever (General disorders) | 52 | 103
Irritability (General disorders) | 71 | 81
Conjunctivitis (Eye disorders) | 6 | 12
Acarodermatitis (Infections and infestations) | 4 | 13
Pneumonia (Infections and infestations) | 54 | 49
Skin infection (Infections and infestations) | 3 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 80 | 80
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 73 | 56
Rash (Skin and subcutaneous tissue disorders) | 1 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.